CLINICAL TRIAL: NCT06183827
Title: Evaluation of Non-Invasive Ventilation/Continuous Positive Airway Pressure for Drowning-related Acute Respiratory Failure
Brief Title: Drowning-related Acute Respiratory Failure
Acronym: CPAPDROWNING
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2023-A01181-44
Record Dates: First submitted 2023-12-05; First posted 2023-12-28 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Drowning
MeSH Terms: conditions — Drowning

STUDY DESIGN:
Intervention Model Description: Multicenter, prospective, cross-over cluster randomized study
Masking Description: Open-label study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the Oxygen Supply strategy (Active Comparator)
  Interventions: Procedure: Emergency Medical Service intervention : Oxygen Supply strategy
- the Continuous Positive Airway Pressure strategy (Experimental)
  Interventions: Procedure: Emergency Medical Service intervention : Continuous Positive Airway Pressure strategy

INTERVENTIONS:
Procedure: Emergency Medical Service intervention : Oxygen Supply strategy — During the 4-month period of control, the care teams will:
  - Use Oxygen Supply by face mask (15Liters/minutes) from pre-hospital to intensive care unit admission until the 6th hour following the start of drowning care (Emergency Medical Service arrival at the scene).
  Indeed, current concepts of advanced prehospital care include the use of oxygen by face mask (15Liters/minutes) and intubation-Mechanical Ventilation in case of failure. The requirement of intubation-Mechanical Ventilation by the Emergency Medical Service (pre-hospital phase) or Intensive Care Unit (hospital phase) practitioners during this first 6 hours period will be left to the discretion of the practitioners in charge of the patient;
  - Continue this strategy in the Intensive Care Unit until the Acute Respiratory Failure resolution allows a reduction of Oxygen Supply. The Oxygen Supply will be reduced progressively litter by litter each 12 hours period with maintenance of capillary saturation up to 92%.
  Arms: the Oxygen Supply strategy
Procedure: Emergency Medical Service intervention : Continuous Positive Airway Pressure strategy — During the 4-month period of experimentation, the care teams will:
  - Use Non-Invasive Ventilation by Continuous Positive Airway Pressure (set between 8 to 10 cm H2O) from pre-hospital setting to Intensive Care Unit admission until the 6th hour following the start of drowning care (Emergency Medical Service arrival at the scene).
  The requirement of Mechanical Ventilation by the Emergency Medical Service (pre-hospital phase) or Intensive Care Unit (hospital phase) practitioners during this first 6 hours period will be left to the discretion of the practitioners in charge of the patient.
  - Continue this strategy in the Intensive Care Unit until the Acute Respiratory Failure resolution allows a reduction of Non-Invasive Ventilation-Continuous Positive Airway Pressure. Non-Invasive Ventilation-Continuous Positive Airway Pressure support will be weaned progressively (left at practitioners' convenience) with maintenance of capillary O2 saturation up to 92%.
  Arms: the Continuous Positive Airway Pressure strategy

SUMMARY:
The purpose of this study is to assess the Non-Invasive Ventilation-Continuous Positive Airway Pressure efficacy (experimental group) for drowning related Acute Respiratory Failure compared to Oxygen Supply by face mask (15Liters/minutes) (control group).

DETAILED DESCRIPTION:
Open-label, multicenter, prospective, cross-over cluster randomized (ratio 1:1), conducted in 16 Emergency Medical Service centers in France :

* Experimental group: Non-Invasive Ventilation-Continuous Positive Airway Pressure (Arm 1)
* Control group: Oxygen Supply by face mask (Arm 2)

Drowning-related acute respiratory failure has important clinical consequences (4 to 18% mortality). No national/international medical consensus exist for its management.

Our team has successively demonstrated that:

* The acute respiratory failure related to drowning in salt or fresh water presented the same clinical pathway and prognosis ;
* Most victims with drowning related acute respiratory failure do no present hemodynamic instability ;
* If the oxygenation is rapidly improved, neurological status is also maintained in acute respiratory failure victims ;
* Pediatric and adult presentations are similar.

Facing an acute respiratory failure, emergency medical service must rapidly choose between oxygen supply by face mask (15 liters /minutes), mechanical ventilation or non-invasive ventilation. mechanical ventilation as non-invasive ventilation present interests and side arms. No comparative study has been conducted between these strategies. The arguments for non-invasive ventilation use specifically in a continuous positive airway pressure mode are:

* Fast recovery of acute respiratory failure in 24h
* Retrospective publications showing that the benefit of non-invasive ventilation probably based on continuous positive airway pressure mode
* Easy implementation of continuous positive airway pressure in the pre-hospital setting (adults, children, newborns)
* Complexity of mechanical ventilation in pre-hospital setting. Our working hypothesis is the efficacy of early use of non-invasive ventilation-continuous positive airway pressure in drowning related acute respiratory failure.

ELIGIBILITY:
Inclusion Criteria:

* Man/boy or woman/girl, 1yo and older.
* Subject suffering from drowning related-Acute Respiratory Failure (whatever the nature of water, salt or fresh) and benefiting from the Emergency Medical Service intervention;
* Acute Respiratory Failure defined as the presence of:

  * Capillary O2 saturation <92% upon Emergency Medical Service first clinical analysis at the drowning scene;
  * Need for oxygen supply 15Liters/minutes to reach capillary O2 saturation ≥ 95%;
  * Combination of Acute Respiratory Failure clinical signs: at least 1 of the following items: respiratory rate >30/min, sternal or clavicular indrawing, abdominal breathing, cyanosis.
* Individual affiliated to or beneficiary of a French health insurance system;
* Individual with the ability to benefit from the two strategies (ambivalence clause);
* Adult Individual having signed written informed consent or child subject with an authorization of the parents.

Exclusion Criteria:

* Individual with hypothermia ≤ 34°C ;
* Individual with neurological distress defined by a Glasgow Coma Scale < 13 at first clinical assessment and during the first 15 minutes of care ;
* Individual with hemodynamic distress defined by a systolic blood tension < 90 mmHg at first clinical assessment and during the first 15 minutes of care ;
* Cardiac arrest or respiratory arrest ;
* Declared pregnancy or breastfeeding ;
* Patient under legal protection regime for adults.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2024-07-24 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Inability to improve oxygen saturation up than 92% | 6 hours
  Indication of intubation/mechanical ventilation requirement in the first 6 hours based on following criteria : Inability to improve oxygen saturation up than 92% despite the ventilatory strategy used;
Glasgow Coma Scale | 6 hours
  Indication of intubation/mechanical ventilation requirement in the first 6 hours based on following criteria : Glasgow Coma Scale < 13
Cardiac arrest occurrence | 6 hours
  Indication of intubation/mechanical ventilation requirement in the first 6 hours based on following criteria : Cardiac arrest occurrence
Systolic arterial pressure | 6 hours
  Indication of intubation/mechanical ventilation requirement in the first 6 hours based on following criteria : Systolic arterial pressure < 90 mmHg
Aspiration | 6 hours
  Indication of intubation/mechanical ventilation requirement in the first 6 hours based on following criteria : Aspiration

CONTACTS AND LOCATIONS:
Locations (9):
- France (9):
  - Centre Hospitalier de la Côte Basque - Urgences, Bayonne
  - Groupe Hospitalier PELLEGRIN - SAMU-SMUR, Bordeaux
  - CH La Rochelle - Urgence, La Rochelle
  - Centre Hospitalier Côte de Lumière - SAMU/SMUR 85, Les Sables-d'Olonne
  - CHU Timone - APHM, Marseille
  - CHU de Montpellier - Hôpital Lapeyronie, Montpellier
  - CHU de Nantes - Urgences/SAMU, Nantes
  - CHU Nice Hôpital Pasteur, Nice
  - CHITS Hôpital Ste Musse, Toulon